CLINICAL TRIAL: NCT06713304
Title: The Effect of a Community-Based Protective Behavioral Strategies Program on Alcohol Use Among Adult Men With Hazardous Alcohol Use in Vietnam
Brief Title: A Community-Based Intervention to Reduce Alcohol Use in Vietnamese Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FONCU2601
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Use
Keywords: Alcohol use; Protective Behavioral Strategies; Adult Men
MeSH Terms: conditions — Alcohol Drinking; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Community-Based Protective Behavioral Strategies Program (Experimental): Participants receive the community-based Protective Behavioral Strategies program
  Interventions: Behavioral: A community-based Protective Behavioral Strategies program
- Control Group (No Intervention): Participants receiving the usual care

INTERVENTIONS:
Behavioral: A community-based Protective Behavioral Strategies program — A 5-week group program delivered in a healthcare setting to teach and practice protective behavioral strategies. The objectives of each session are:
  Session 1: Setting Safe Drinking Limit: The participants can identify the risk related to their drinking behavior, calculate a standard drink, and set a safe drinking limit.
  Session 2: Choosing Nonalcoholic Drinks: The participants can understand the benefits of using nonalcoholic beverages and identify and select nonalcoholic beverages.
  Session 3: Planning Ahead: The participants can make a plan to stop using during drinking events and know how to say "no" to alcohol use.
  Session 4: Slowing down drinking: The participants can understand the benefits of slowing down drinking and know how to slow down their drinks.
  Session 5: Avoid Risky Drinking Situations: The participants can understand the negative effects of excessive drinking and know how to avoid excessive drinking.
  Arms: A Community-Based Protective Behavioral Strategies Program

SUMMARY:
This study aims to evaluate the effectiveness of a community-based Protective Behavioral Strategies (PBS) program in reducing alcohol use, severity of alcohol-related problems, and intention to use alcohol among people with hazardous alcohol use (HAU) in Vietnam. In this randomized controlled trial, 104 men aged 35-44 years, identified as having HAU (Alcohol Use Disorders Identification Test score = 8-15), will be recruited from a rural area in Thai Nguyen province, Vietnam. Participants will be randomly assigned in a 1:1 ratio to either the intervention or control group using stratified blocked randomization. The intervention group will participate in a community-based PBS program, which includes five weekly 90-minute sessions, with Short Message Service (SMS) reminders sent three times weekly after each session to reinforce PBS practices. The control group will receive usual care only.

The primary outcome is alcohol use, assessing both the quantity and frequency of consumption, measured at 1 month and 3 months post-intervention. Secondary outcomes include the severity of alcohol-related problems and intention to use alcohol. These will be assessed at baseline and the 3-month follow-up. Two-way repeated measures Multivariate analysis of variance (MANOVA) and regression models will be conducted to evaluate the effects of the intervention on the primary and secondary outcomes.

DETAILED DESCRIPTION:
* Background and significance: Hazardous alcohol use (HAU) represents a significant public health concern, particularly among adult men in Vietnam. Effective interventions are needed to reduce HAU and its associated health risks. Protective Behavioral Strategies (PBS) have shown promise in mitigating HAU behaviors by promoting safer drinking practices and enhancing self-regulation among individuals.

* Study objectives:

  1. To compare the differences in the primary outcome (alcohol use) between the intervention and control groups at 1 month and 3 months post-intervention, and the differences in the secondary outcomes (severity of alcohol-related problems and intention to use alcohol) at 3 months post-intervention.
  2. To compare the differences in the primary outcome (alcohol use) at 1 month and 3 months post-intervention, and the differences in the secondary outcomes (severity of alcohol-related problems and intention to use alcohol) at 3 months post-intervention, within the intervention group compared to the pre-test.
* Study design:

This study employs a randomized controlled design. Alcohol use will be measured at both 1 month and 3 months after the intervention, whereas the secondary outcomes will be measured at 3 months. The 1-month follow-up allows for the evaluation of immediate changes in drinking behavior, while the 3-month follow-up assesses whether these changes are sustained. By comparing outcomes across both time points, the study can track the trajectory of the intervention's impact and identify any patterns of relapse or continued improvement. These follow-up periods align with common practice in alcohol intervention research.

* Intervention: The intervention group will participate in a community-based PBS program, which is structured around PBS as its central framework, enhanced by Alcohol Brief Intervention (functioning as a motivating component), and Behavioral Skills Training model (enhancing the learning of each PBS skill through a structured approach: instruction, modeling, rehearsal, and feedback). The community-based PBS program consists of 5 weekly sessions including Setting safe drinking limits, Choosing non-alcoholic drinks, Planning Ahead, Slowing down drinking, and Avoiding Risky Drinking situations each lasting 90 minutes.

The sessions will be delivered by the researcher in an in-person group format (10-12 participants per group) at a healthcare facility. Each session is structured as follows: Part 1-30 minutes: Introduction, relationship-building, and reviewing previous content. This segment focuses on fostering a supportive environment and reinforcing participants' connection with the program. Part 2-60 minutes: Learning and practicing PBS. Participants will be introduced to specific strategies each week, followed by hands-on practice, group discussions, and scenario-based exercises that encourage the application of PBS in real-life situations.

After each session, participants will receive three Short Message Service (SMS) text messages per week (a random day, Friday, and Saturday). These messages encourage participants to apply the PBS learned in the group sessions. The main activities in each session are briefly summarized below.

* Usual care: Usual care refers to the standard services provided by primary care nurses to people with HAU in the community, as per national guidelines. This typically includes educational sessions on the adverse effects of alcohol, guidance on relevant laws and health regulations, and referrals to healthcare services.

* Outcome measures:

  * Alcohol use is measured by both the amount and frequency of alcohol consumption. The amount of alcohol use is quantified as the total grams of pure alcohol that participants consumed per week in the previous month measuring at baseline, 1 month, and 3 months post-intervention. This is calculated using the formula: Volume (ml) × Alcohol by Volume (%) × 0.79, where Alcohol by Volume is the alcohol by volume percentage and 0.79 is the conversion factor for the density of ethanol (Vietnamese Ministry of Health, 2020). Frequency of alcohol use is defined as the number of days per week in the previous month that participants consume alcohol measuring at baseline, 1 month, and 3 months post-intervention. These variables are measured using the Alcohol Timeline Follow back.
  * The severity of alcohol-related problems refers to the participants' self-report of the extent and intensity of negative consequences resulting from alcohol use, measured at baseline and 3 months post-intervention. These consequences are categorized into physical, intrapersonal, interpersonal, social responsibility, and impulse control domains. This variable is measured using the Drinker Inventory of Consequences.
  * Intention to use alcohol is operationally defined as participants' self-reported intention or willingness to consume alcohol within the next 30 days. This is measured using a 7-point Likert scale at baseline and 3 months post-intervention in response to the statement: "I intend to drink alcohol in the next 30 days" with responses ranging from 1 to 7.
* Data Analysis:

Data will be analyzed using Statistical Package for the Social Sciences (SPSS) version 28.0. Two-way repeated measures Multivariate analysis of variance (MANOVA) will be employed to assess changes in outcomes over time and between groups. Regression models will be utilized to explore the relationship between the intervention and changes in alcohol use and associated outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Having a total AUDIT score from 8 to 15
* Completing at least primary school
* Able to use the Vietnamese language
* Having a mobile phone
* Willing to participate in this study

Exclusion Criteria:

* Using alcohol and other illicit drugs at the same time
* Having any physical illness or psychiatric disorders

Ages: 35 Years to 44 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 104 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Alcohol use | Baseline, 1 month and 3 months post-intervention
  Alcohol use is measured by both the amount and frequency of alcohol consumption. The amount of alcohol use is quantified as the total grams of pure alcohol that participants consumed per week in the previous month measuring at baseline, 1 month, and 3 months post-intervention. This is calculated using the formula: Volume (ml) × ABV(%) × 0.79, where ABV is the alcohol by volume percentage and 0.79 is the conversion factor for the density of ethanol. Frequency of alcohol use is defined as the number of days per week in the previous month that participants consume alcohol measuring at baseline, 1 month, and 3 months post-intervention. These variables are measured using the Alcohol Timeline Follow back (TLFB).

SECONDARY OUTCOMES:
Severity of alcohol-related problems | Baseline and 3 months post-intervention
  The severity of alcohol-related problems refers to the participants' self-report of the extent and intensity of negative consequences resulting from alcohol use, measured at baseline and 3 months post-intervention. These consequences are categorized into physical, intrapersonal, interpersonal, social responsibility, and impulse control domains. This variable is measured using the Drinker Inventory of Consequences (DrInC).
Intention to use alcohol | Baseline and 3 months post-intervention
  Intention to use alcohol is operationally defined as participants' self-reported intention or willingness to consume alcohol within the next 30 days. This is measured using a 7-point Likert scale at baseline and 3 months post-intervention in response to the statement: "I intend to drink alcohol in the next 30 days" with responses ranging from 1 to 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn University, Faculty of Nursing, Bangkok, Bangkok, Thailand, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: the IPD and supporting information will be available 6 months after the publication of primary results and will remain accessible for 2 years.
Access Criteria: Researchers with a valid scientific purpose may access the de-identified IPD and supporting information upon submission of a data-sharing request. Requests should include a research proposal and the intended use of the data.